CLINICAL TRIAL: NCT03690960
Title: Evaluation of the Antimicrobial Effect of Pre-synthesized Novel Antibiotic Electrospun Nanofibers as an Intracanal Delivery Strategy for Regenerative Endodontics A Randomized Clinical Trial
Brief Title: Antimicrobial Effect of Modified Antibiotic Nanofibers for Regenerative Endodontics Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, sara Gamal Ahmed, Ass.lecturer of endodotics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cairo University dentistry
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Necrosis, Pulp
Keywords: immature teeth
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- electrospun TAP nanofibers (Experimental): Revascularization procedure with Electrospun TAP nanofibers as as an intracanal medicament for immature necrotic teeth
  Interventions: Procedure: electrospun TAP nanofibers
- modified TAP paste (Active Comparator): Revascularization procedure with modified TAP paste as an intracanal medicament for immature necrotic teeth
  Interventions: Procedure: modified TAP paste

INTERVENTIONS:
Procedure: electrospun TAP nanofibers — electrospun TAP loaded nanofibers containing modified triple antibiotic paste of clindamycin , ciprofloxacin and metronidazole by electrospinning process will be placed in the root canals. The access cavity will be sealed with temporary filling material
  Arms: electrospun TAP nanofibers
Procedure: modified TAP paste — modified TAP paste will be prepared by mixing equal proportions of CIP, MET and CLIN then placed inside the root canal, access cavity will be sealed with temporary filling
  Arms: modified TAP paste

SUMMARY:
The treatment for immature teeth with pulp necrosis can be carried out through apexification or regenerative endodontics procedures including platelet rich plasma (PRP), platelet rich fibrin (PRF) and injectable PRF, these techniques used alone or in combination. Revascularization therapy carries on more advantages than apexification, such as inducing root-end development and reinforcement. However, apical repair will not happen in the presence of inflamed and infected tissue.the aim of this study is to evaluate the antimicrobial effect of pre-synthesized novel antibiotic loaded electrospun nanofibers used in patients with immature necrotic teeth.

DETAILED DESCRIPTION:
Title: Evaluation of the Antimicrobial Effect of Pre-synthesized Novel Antibiotic Electrospun Nanofibers as an Intracanal Delivery Strategy for Regenerative Endodontics - A Randomized Clinical Trial

Rationale Regenerative endodontics technique outcome depends on microbial elimination because apical repair will not happen in the presence of infected tissues. It is well established that bacteria are essential for the development of pulpal and periapical pathosis. Eradication or control of bacteria may provide optimal treatment outcome. However, elimination of bacteria from infected root canal systems is challenging. Numerous measures have been described to reduce the number of bacteria in the root canal system, including the use of various instrumentation techniques, irrigation regimens and intra-canal medicaments. There is no definitive evidence in the literature that all these measures result in a bacteria-free root canal system.

Therefore additional methods such as the use of intra-canal medicaments are required in order to maximize disinfection of root canal system and kill as many bacteria as possible. Antibiotics have been proposed as intracanal medicament but any single antibiotic is unlikely effective to sterilize diverse flora in root canal infection.

Recently, triple antibiotic mixture (TAP) has been reported for successful disinfection of infected root dentine. This mixture consist of ciprofloxacin (CIP), metronidazole (MET) and minocycline (MINO) which consistently sterilize bacteria of infected dentine and infected pulps . Specifically, MET is a bactericidal imidazole that is highly effective against obligate anaerobic bacteria, CIP is a bactericidal broad-spectrum synthetic quinolone and MINO is a bacteriostatic broad-spectrum tetracycline.

However, as minocycline binds to dentin and causes tooth discoloration, it is recommended to remove minocycline from TAP and use only MET and CIP, or to use modified TAPs containing cefaclor or clindamycin (CLIN). CLIN is a bacteriostatic lincosamide known for its efficacy against a broad spectrum of endodontic bacteria.

In recent years, an innovative strategy has been considered to develop a low-concentration, yet antimicrobially effective and biocompatible polymer-based nanofibrous electrospun scaffolds as a drug delivery system to promote intracanal biofilm eradication . Electrospinning has been considered as a highly effective process to obtain extracellular matrix (ECM) mimicking structures with adequate chemistry and three-dimensional porous architectures Moreover, it has enabled the synthesis of bioactive nanofibrous scaffolds The electrospinning technology has attracted great interest in recent decades, thanks to its capability of easily and effectively processing a huge range of polymeric materials in form of nanofibers. In recent years, the health concerns associated with the systemic side effects of synthetic compounds used in medicine and the emergence of antibiotic resistance of pathogens have driven electrospinning research towards the development of antibiotic loaded nanofibers.

Hypothesis To test the null hypothesis, which is in patients with necrotic immature teeth, will the use of pre-synthesized clindamycin modified triple antibiotic electrospun nanofibers have more profound antimicrobial effect than modified triple antibiotic paste.

Objectives of the present study

* Primary objective To compare the antimicrobial effect of pre-synthesized novel antibiotic loaded nanofibers used in patients with immature necrotic teeth with modified triple antibiotic paste.
* Secondary objective To evaluate the morphology of pre-synthesized antibiotic loaded electrospun nanofibers.

ELIGIBILITY:
Inclusion Criteria:

Maxillary or mandibular single-root tooth with:

* Non-vital response of pulp tissue.
* Immature root.
* Asymptomatic patients.

Exclusion Criteria:

1. Patients allergic to metronidazole, ciprofloxacin, or clindamycin to avoid allergic reaction in the intervention group.
2. Patients who received antibiotics in the past 3 months.
3. Vital cases or previously accessed teeth.
4. Teeth with unfavorable conditions for rubber-dam application.
5. Patients with systemic and immune-compromising disease as they have impaired healing

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
antimicrobial effect | 2-3 weeks
  number of colony forming units of bacteria after using the intracanal medicaments

SECONDARY OUTCOMES:
morphology of nanofibers | 1 week
  surface morphology will be studied under the scanning electron microscope